CLINICAL TRIAL: NCT01414296
Title: Extended 39-Week Study of PSMA ADC Following the Initial 12-Week Dose-escalation Study in Subjects With Progressive, Castration-resistant, Metastatic Prostate Cancer
Brief Title: Extended Study of Prostate-specific Membrane Antigen Antibody-Drug Conjugate in Subjects With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSMA ADC 1301EXT
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PSMA ADC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: PSMA ADC

INTERVENTIONS:
Drug: PSMA ADC — PSMA ADC administered IV

SUMMARY:
Prostate-specific Membrane Antigen Antibody-Drug Conjugate (PSMA ADC) 1301EXT is an open-label, nonrandomized, phase 1 extension study of PSMA ADC administered IV in subjects with progressive CMPC that has progressed after prior taxane therapy. Subjects who have participated in PSMA ADC 1301 and who, in the opinion of the PI, are likely to benefit from continued treatment with PSMA ADC will be enrolled in PSMA ADC 1301EXT.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have completed the PSMA ADC 1301 study and who, in the opinion of the investigator, have derived benefit from treatment with PSMA ADC.
2. A diagnosis of progressive, castration-resistant, metastatic prostate cancer.
3. Prior chemotherapy regimens, one of which contains taxane.
4. Eastern Cooperative Oncology Group status of 0 or 1

Exclusion Criteria:

1. Clinically significant cardiac disease or severe debilitation pulmonary disease
2. Evidence of an active infection requiring ongoing antibiotic therapy
3. History of drug and/or alcohol abuse

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-01; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events | 39 weeks
  Safety and tolerability of PSMA ADC as measured by all adverse events, hematology, blood chemistry, and urine values, vital signs, electrocardiogram, and physical exam.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Israel, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States